CLINICAL TRIAL: NCT06101849
Title: Evaluating an Online Interprofessional Chronic Pain Management Group for Survivors of Breast Cancer: A Feasibility Study of a Randomized Controlled Trial
Brief Title: Chronic Cancer Pain Management Program
Acronym: ICMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Karen Zhang, Clinical, Health and Rehabilitation Psychologist, Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16187
Record Dates: First submitted 2023-09-28; First posted 2023-10-26 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Cancer, Treatment-Related; Pain Cancer
Keywords: Pain; Breast Cancer; Cancer Pain; Pain Management; psycho-oncology; Psychology; quality of life
MeSH Terms: conditions — Breast Neoplasms; Neoplasms, Second Primary; Cancer Pain; Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: A pre-post study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer Pain Management Group (Experimental): Participants in the study will attend a 6-week online pain management program (I-Can-Manage-Pain after cancer) that will cover the topics of understanding cancer pain, exercises to manage pain and psychological strategies to cope with pain. Questionnaires will be administered before and after the program
  Interventions: Behavioral: I-Can-Manage-Pain after cancer (Pain Management Program)

INTERVENTIONS:
Behavioral: I-Can-Manage-Pain after cancer (Pain Management Program) — 6-week online interprofessional cancer pain management program (I-Can-Manage-Pain after cancer) for survivors of breast cancer. The program will cover the topics of understanding cancer pain, exercises to manage pain and psychological strategies to cope with pain

SUMMARY:
The goal of this research study is to evaluate an online inter-professional pain management program for survivors of breast cancer.

The main questions it aims to answer:

1. whether this treatment will help address the pain management concerns of patients,
2. whether it is feasible to offer this treatment in the future as multi-centre randomized controlled trial (RCT).

Participants will be asked to attend a 6-week online pain management group sessions (1h/week). Participants will also be asked to fill out questionnaires before and after the program completion.

DETAILED DESCRIPTION:
Survivors of breast cancer often experience chronic pain that is undertreated and gets in the way of their functioning, relationships, mental health, and quality of life. There is little research on the best ways of treating chronic pain in cancer that make good use of all the expertise offered by different health care providers such as nurses, psychologists, and physiotherapists. In addition, little is known about how to offer such a service in an online format.

This study aims to pilot an online interprofessional pain management program for survivors of breast cancer. The investigators would like to know whether this treatment will help address the pain management concerns of patients, and whether it is feasible to offer this treatment in the future as multi-centre randomized controlled trial (RCT).

Participants in the study will attend a 6-week online pain management program (I-Can-Manage-Pain after cancer) that will cover the topics of understanding cancer pain, exercises to manage pain and psychological strategies to cope with pain. Questionnaires will be administered before and after the program to assess their satisfaction and changes in outcomes related to pain, quality of life, confidence to manage their pain, and use of health care services. The feasibility of implementing the study and the program will be pre-determined by an acceptability criteria for patient recruitment, completion of questionnaires, participation in the online sessions, and satisfaction with the pain management program.

It is hoped that study findings will help inform the development of treatment programs to improve post-treatment pain management and the quality of life of survivors of breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of Stage 1-3 breast cancer;
2. had surgical excision at least 3 months ago;
3. completed neoadjuvant/adjuvant chemotherapy and/or radiation treatment at least 4 months ago;
4. within 5 years post active cancer treatment;
5. persistent pain within the last 3 months that is bothersome;
6. medical clearance to participate in the intervention
7. over 18 years of age;
8. verbal fluency in English;
9. have access to internet and technology to participate in the online program. Patients currently receiving adjuvant endocrine therapy or molecularly targeted therapies or who have completed these therapies within the last 5 years are eligible to participate.

Exclusion Criteria:

* Participants will be excluded from the study if they:

  1. demonstrate significant cognitive impairment as determined by the clinical judgment of the provider;
  2. have a pre-existing non-cancer pain condition,
  3. have severe emotional distress that interferes with group participation as determined by scores above 15 on the Patient Health Questionnaire-9.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Pain Interference. | 6 weeks
  This construct will be measured using the 6-item Patient-Reported Outcome Measurement Information System (PROMIS) Pain Interference Scale. (PIS) The PIS uses a 5-point rating scale to determine the degree to which an individual perceives their pain symptoms to interfere with their physical, mental and social functioning. Sum of raw scores will be translated to a T-score using a conversion table. A T-score of 50 with a standard deviation of 10 is the average for the general population based on United States Data. The minimally important difference20 for the PIS scores among pain samples ranges from 2 to 3 T-score points.

SECONDARY OUTCOMES:
Pain intensity. | 6 weeks
  The three-item PROMIS Pain Intensity-Short Form measures the severity of pain over a course of 7 days. Scores on this scale range from 3-15. Higher scores indicate higher pain intensity
Pain Catastrophizing; | 6 weeks
  Catastrophizing is the anticipation of negative pain experience and will be measured using the 13-item Pain Catastrophizing Scale. The scores on this scale range from 0-52 and higher scores indicate higher tendency for pain catastrophizing
Psychological Distress (depression, anxiety, stress) | 6 weeks
  Will be assessed by degree of depression, anxiety, stress. The 21-item Depression, Anxiety and Stress Scale (DASS-21) will be used to measure mood, anxiety and stress symptoms over the past week. Higher scores on the three subscales of depression, anxiety and stress indicate higher emotional distress.
Psychological Distress (Fear of Cancer recurrence) | 6 weeks
  Fear of cancer recurrence will be assessed using the 6-item Cancer Worry Scale (CWS). Score of 14 or above indicates high levels of fear of recurrence
Self-Efficacy | 6 weeks
  Will be assessed using the brief version of the cancer behavior inventory (CBI-B). The CBI is a 12-item measure examines the degree to which an individual feels confident in self-managing their cancer. This measure shows good internal consistency. Higher scores indicator greater confidence in self-managing cancer.
Healthcare Utilization | 6 weeks
  Will be assessed using the Health Service Utilization Questionnaire. This questionnaire assesses health care facility visits, procedures obtained and support services used. Higher numbers indicates more usage of healthcare services
Patient Satisfaction | 6 weeks
  Items 12-14 on the Patient Satisfaction Survey will be used to measure the extent to which patients understood the survey questions, and their satisfaction with the survey length
Trial adherence and fidelity | 12 months
  Percentage of participants completing the trial questionnaire and the intervention program.
Trial Feasibility (ability to recruit patients) | 12 months
  ability to recruit patients will be assessed using the trial screening and recruitment log. A recruitment of 1-2 participants per week is considered sufficient.
Patients' satisfaction with the intervention. | 12 months
  patients' satisfaction with the intervention will be measured using the patients' satisfaction survey (PSS). Scores on items 1-4 and 10-14 of PSS range between 1-5. Higher scores on items 1-4 and 10-14 indicates higher satisfaction. Other items will be analyzed qualitatively.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Zhang, PHD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Int J Nurs Stud. 2013 May;50(5):587-92. doi: 10.1016/j.ijnurstu.2012.09.010. Epub 2012 Nov 15. No abstract available. PMID 23159157
- [Background] Orsmond GI, Cohn ES. The Distinctive Features of a Feasibility Study: Objectives and Guiding Questions. OTJR (Thorofare N J). 2015 Jul;35(3):169-77. doi: 10.1177/1539449215578649. PMID 26594739
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Burckhardt CS, Jones KD. Effects of chronic widespread pain on the health status and quality of life of women after breast cancer surgery. Health Qual Life Outcomes. 2005 Apr 28;3:30. doi: 10.1186/1477-7525-3-30. PMID 15860132
- [Background] Hamood R, Hamood H, Merhasin I, Keinan-Boker L. Chronic pain and other symptoms among breast cancer survivors: prevalence, predictors, and effects on quality of life. Breast Cancer Res Treat. 2018 Jan;167(1):157-169. doi: 10.1007/s10549-017-4485-0. Epub 2017 Aug 31. PMID 28861642
- [Background] Classification of chronic pain. Descriptions of chronic pain syndromes and definitions of pain terms. Prepared by the International Association for the Study of Pain, Subcommittee on Taxonomy. Pain Suppl. 1986;3:S1-226. No abstract available. PMID 3461421
- [Background] Feeney LR, Tormey SM, Harmon DC. Breast cancer and chronic pain: a mixed methods review. Ir J Med Sci. 2018 Nov;187(4):877-885. doi: 10.1007/s11845-018-1760-y. Epub 2018 Feb 5. PMID 29404844
- [Background] Wang K, Yee C, Tam S, Drost L, Chan S, Zaki P, Rico V, Ariello K, Dasios M, Lam H, DeAngelis C, Chow E. Prevalence of pain in patients with breast cancer post-treatment: A systematic review. Breast. 2018 Dec;42:113-127. doi: 10.1016/j.breast.2018.08.105. Epub 2018 Sep 4. PMID 30243159
- [Background] Forsythe LP, Alfano CM, George SM, McTiernan A, Baumgartner KB, Bernstein L, Ballard-Barbash R. Pain in long-term breast cancer survivors: the role of body mass index, physical activity, and sedentary behavior. Breast Cancer Res Treat. 2013 Jan;137(2):617-30. doi: 10.1007/s10549-012-2335-7. Epub 2012 Dec 15. PMID 23242613
- [Background] Vilholm OJ, Cold S, Rasmussen L, Sindrup SH. The postmastectomy pain syndrome: an epidemiological study on the prevalence of chronic pain after surgery for breast cancer. Br J Cancer. 2008 Aug 19;99(4):604-10. doi: 10.1038/sj.bjc.6604534. PMID 18682712
- [Background] Levy MH, Chwistek M, Mehta RS. Management of chronic pain in cancer survivors. Cancer J. 2008 Nov-Dec;14(6):401-9. doi: 10.1097/PPO.0b013e31818f5aa7. PMID 19060605
- [Background] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Background] Novy DM, Aigner CJ. The biopsychosocial model in cancer pain. Curr Opin Support Palliat Care. 2014 Jun;8(2):117-23. doi: 10.1097/SPC.0000000000000046. PMID 24690764
- [Background] Paice JA, Portenoy R, Lacchetti C, Campbell T, Cheville A, Citron M, Constine LS, Cooper A, Glare P, Keefe F, Koyyalagunta L, Levy M, Miaskowski C, Otis-Green S, Sloan P, Bruera E. Management of Chronic Pain in Survivors of Adult Cancers: American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2016 Sep 20;34(27):3325-45. doi: 10.1200/JCO.2016.68.5206. Epub 2016 Jul 25. PMID 27458286
- [Background] McCowat M, Fleming L, Vibholm J, Dixon D. The Psychological Predictors of Acute and Chronic Pain in Women Following Breast Cancer Surgery: A Systematic Review. Clin J Pain. 2019 Mar;35(3):261-271. doi: 10.1097/AJP.0000000000000672. PMID 30531400
- [Background] Glare PA, Davies PS, Finlay E, Gulati A, Lemanne D, Moryl N, Oeffinger KC, Paice JA, Stubblefield MD, Syrjala KL. Pain in cancer survivors. J Clin Oncol. 2014 Jun 1;32(16):1739-47. doi: 10.1200/JCO.2013.52.4629. Epub 2014 May 5. PMID 24799477
- [Background] Chen CX, Kroenke K, Stump TE, Kean J, Carpenter JS, Krebs EE, Bair MJ, Damush TM, Monahan PO. Estimating minimally important differences for the PROMIS pain interference scales: results from 3 randomized clinical trials. Pain. 2018 Apr;159(4):775-782. doi: 10.1097/j.pain.0000000000001121. PMID 29200181
- [Background] Miller KD, Siegel RL, Lin CC, Mariotto AB, Kramer JL, Rowland JH, Stein KD, Alteri R, Jemal A. Cancer treatment and survivorship statistics, 2016. CA Cancer J Clin. 2016 Jul;66(4):271-89. doi: 10.3322/caac.21349. Epub 2016 Jun 2. PMID 27253694
- [Background] Sheinfeld Gorin S, Krebs P, Badr H, Janke EA, Jim HS, Spring B, Mohr DC, Berendsen MA, Jacobsen PB. Meta-analysis of psychosocial interventions to reduce pain in patients with cancer. J Clin Oncol. 2012 Feb 10;30(5):539-47. doi: 10.1200/JCO.2011.37.0437. Epub 2012 Jan 17. PMID 22253460
- [Background] Johannsen M, Farver I, Beck N, Zachariae R. The efficacy of psychosocial intervention for pain in breast cancer patients and survivors: a systematic review and meta-analysis. Breast Cancer Res Treat. 2013 Apr;138(3):675-90. doi: 10.1007/s10549-013-2503-4. Epub 2013 Apr 4. PMID 23553565
- [Background] Syrjala KL, Donaldson GW, Davis MW, Kippes ME, Carr JE. Relaxation and imagery and cognitive-behavioral training reduce pain during cancer treatment: a controlled clinical trial. Pain. 1995 Nov;63(2):189-198. doi: 10.1016/0304-3959(95)00039-U. PMID 8628584
- [Background] Syrjala KL, Jensen MP, Mendoza ME, Yi JC, Fisher HM, Keefe FJ. Psychological and behavioral approaches to cancer pain management. J Clin Oncol. 2014 Jun 1;32(16):1703-11. doi: 10.1200/JCO.2013.54.4825. Epub 2014 May 5. PMID 24799497
- [Background] Heathcote LC, Eccleston C. Pain and cancer survival: a cognitive-affective model of symptom appraisal and the uncertain threat of disease recurrence. Pain. 2017 Jul;158(7):1187-1191. doi: 10.1097/j.pain.0000000000000872. No abstract available. PMID 28195857
- [Background] Gilbody S, Richards D, Brealey S, Hewitt C. Screening for depression in medical settings with the Patient Health Questionnaire (PHQ): a diagnostic meta-analysis. J Gen Intern Med. 2007 Nov;22(11):1596-602. doi: 10.1007/s11606-007-0333-y. Epub 2007 Sep 14. PMID 17874169
- [Background] Arain M, Campbell MJ, Cooper CL, Lancaster GA. What is a pilot or feasibility study? A review of current practice and editorial policy. BMC Med Res Methodol. 2010 Jul 16;10:67. doi: 10.1186/1471-2288-10-67. PMID 20637084
- [Background] Katz L, Patterson L, Zacharias R. Evaluation of an interdisciplinary chronic pain program and predictors of readiness for change. Can J Pain. 2019 Apr 12;3(1):70-78. doi: 10.1080/24740527.2019.1582296. eCollection 2019. PMID 35005395
- [Background] Borrelli B. The Assessment, Monitoring, and Enhancement of Treatment Fidelity In Public Health Clinical Trials. J Public Health Dent. 2011 Winter;71(s1):S52-S63. doi: 10.1111/j.1752-7325.2011.00233.x. PMID 21499543
- [Background] Tariman JD, Berry DL, Halpenny B, Wolpin S, Schepp K. Validation and testing of the Acceptability E-scale for web-based patient-reported outcomes in cancer care. Appl Nurs Res. 2011 Feb;24(1):53-8. doi: 10.1016/j.apnr.2009.04.003. Epub 2009 Sep 18. PMID 20974066
- [Background] Vaismoradi M, Turunen H, Bondas T. Content analysis and thematic analysis: Implications for conducting a qualitative descriptive study. Nurs Health Sci. 2013 Sep;15(3):398-405. doi: 10.1111/nhs.12048. Epub 2013 Mar 11. PMID 23480423
- [Background] Cook KF, Jensen SE, Schalet BD, Beaumont JL, Amtmann D, Czajkowski S, Dewalt DA, Fries JF, Pilkonis PA, Reeve BB, Stone AA, Weinfurt KP, Cella D. PROMIS measures of pain, fatigue, negative affect, physical function, and social function demonstrated clinical validity across a range of chronic conditions. J Clin Epidemiol. 2016 May;73:89-102. doi: 10.1016/j.jclinepi.2015.08.038. Epub 2016 Mar 4. PMID 26952842
- [Background] Askew RL, Cook KF, Revicki DA, Cella D, Amtmann D. Evidence from diverse clinical populations supported clinical validity of PROMIS pain interference and pain behavior. J Clin Epidemiol. 2016 May;73:103-11. doi: 10.1016/j.jclinepi.2015.08.035. Epub 2016 Feb 27. PMID 26931296
- [Background] Douma KF, Aaronson NK, Vasen HF, Gerritsma MA, Gundy CM, Janssen EP, Vriends AH, Cats A, Verhoef S, Bleiker EM. Psychological distress and use of psychosocial support in familial adenomatous polyposis. Psychooncology. 2010 Mar;19(3):289-98. doi: 10.1002/pon.1570. PMID 19382100
- [Background] Heitzmann CA, Merluzzi TV, Jean-Pierre P, Roscoe JA, Kirsh KL, Passik SD. Assessing self-efficacy for coping with cancer: development and psychometric analysis of the brief version of the Cancer Behavior Inventory (CBI-B). Psychooncology. 2011 Mar;20(3):302-12. doi: 10.1002/pon.1735. PMID 20878830
- [Background] Groenvold M, Petersen MA, Aaronson NK, Arraras JI, Blazeby JM, Bottomley A, Fayers PM, de Graeff A, Hammerlid E, Kaasa S, Sprangers MA, Bjorner JB. EORTC QLQ-C15-PAL: the new standard in the assessment of health-related quality of life in advanced cancer? Palliat Med. 2006 Mar;20(2):59-61. doi: 10.1191/0269216306pm1133xx. No abstract available. PMID 16613400
- [Background] Sullivan, M. J. L., Bishop, S. R., & Pivik, J. (1995). The Pain Catastrophizing Scale: Development and validation. Psychological Assessment, 7(4), 524-532. https://doi.org/10.1037/1040-3590.7.4.524
- [Background] Lovibond, S.H. & Lovibond, P.F. (1995). Manual for the Depression Anxiety Stress Scales. (2nd. Ed.) Sydney: Psychology Foundation.
- [Background] Canadian Pain Task Force. (June, 2019). Chronic pain in Canada: Laying a foundation for action.https://www.canada.ca/content/dam/hc-sc/documents/corporate/about-health-canada/publicengagement/external-advisory-bodies/canadian-pain-task-force/report-2019/canadian-pain-task-forceJune-2019-report-en.pdf
- [Background] Cancer Care Ontario. (April, 2012). Cancer-related pain management. Cancer Care Ontario: Toronto, ON.
- [Background] The British Pain Society. (November 2013). Guidelines for pain management programmes for adults: An evidence-based review prepared on behalf of the British Pain Society. https://www.britishpainsociety.org/static/uploads/resources/files/pmp2013_main_FINAL_v6.pdf